CLINICAL TRIAL: NCT06513195
Title: Endoscopic Ultrasound Guided Response Assessment to Non-selective Beta-blockers in the Treatment of Clinically Significant Portal Hypertension
Brief Title: EUS-guided Response Assessment to NSBB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: s67433
Record Dates: First submitted 2024-07-08; First posted 2024-07-22 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2023-12

CONDITIONS: Portal Hypertension Related to Cirrhosis
Keywords: portal hypertension; EUS-PPG; HVPG; cirrhosis; non-selective beta blockers
MeSH Terms: conditions — Hypertension, Portal; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EUS-PPG before and after NSBB (Experimental): Patients will undergo EUS-PPG and HVPG before and after NSBB treatment and will thus serve as their own control.
  Interventions: Procedure: endoscopic ultrasound-guided portal pressure measurement

INTERVENTIONS:
Procedure: endoscopic ultrasound-guided portal pressure measurement — The portal pressure gradient will be determined by endoscopic ultrasound-guided pressure measurement in the hepatic vein and the portal vein. The gradient will be calculated by substracting the hepatic vein pressure from the portal vein pressure.
  Other Names: EUS-PPG

SUMMARY:
The goal of this clinical trial is to learn if endoscopic ultrasound (EUS)-guided portal pressure measurement can determine the treatment response to non-selective beta-blockers (NSBB) in patients with cirrhosis and clinically significant portal hypertension (CSPH). Participants will undergo EUS-guided portal pressure measurement before start of Carvedilol en after three months of treatment. EUS-guided measurements will be paired with transjugular hepatic venous pressure gradient (HVPG) measurement as well as non-invasive tests for assessment of portal hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical and/or pathological diagnosis of compensated cirrhosis.
* Patients with suspicion of CSPH and thus indication for NSBB treatment.
* Patients not yet on NSBB therapy.
* Patients willing and able to undergo repeated HVPG and EUS-guided pressure measurements as per protocol.

Exclusion Criteria:

General criteria

* Patient is <18 or >80 years of age
* Patient is pregnant, breast-feeding or planning to become pregnant during the course of the study
* Patient is unwilling or unable to sign the informed consent
* Patients in whom general anesthesia or endoscopic procedures are contraindicated Medical criteria
* Patients with cirrhosis and HCC Portopulmonary hypertension Portal or splanchnic venous thrombosis Prior TIPS Prior liver transplantation
* Non-cirrhotic portal hypertension or pre-sinusoidal liver disease
* Cholestatic liver disease with total bilirubin >3 mg/dl
* Previous total or partial splenectomy
* Known infection that is not controlled by medical intervention
* Patients with contraindications for non-selective beta-blocker therapy, including but not limited to the following baseline vital signs:

Systolic BP <100 mmHg HR <50 bpm

* Patients with reduced life expectancy described by an ASA score of 4 or 5
* INR >1.7 or platelet count <50.000 per mm3
* eGFR <50 ml/min/1.73m2 (CKD-EPI formula) Anatomical criteria
* Anatomical abnormalities that prevent access via EUS-guided puncture to the hepatic vein or intrahepatic portion of the portal vein, including anatomy that predisposes to difficult to reach puncture sites or an inadequate needle angle.
* Visualization of ascites interposing the puncture tract on EUS
* Diagnosis of portal vein thrombosis during EUS
* Evidence of active gastrointestinal bleeding during EUS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
EUS-guided response assessment to NSBB in the treatment of CSPH. | Three months
  To assess if a positive response to non-selective beta-blockers (NSBB) treatment, as determined by a reduction of 10% or more in the hepatic venous pressure gradient (HVPG) and/or a decrease to values less than 12 mmHg, can be similarly observed using endoscopic ultrasound-guided portal pressure gradient (EUS-PPG) measurement.

SECONDARY OUTCOMES:
Correlation of EUS-PPG with HVPG | Three months
  To assess the correlation of EUS-PPG and HVPG before treatment start as well as after treatment start with NSBB
Correlation of FHVP with HVP. | Three months
  To assess the correlation of EUS-guided hepatic venous pressure (HVP) and transjugular free hepatic venous pressure (FHVP) measurement before treatment start as well as after treatment start with NSBB.
Correlation of PVP with WHVP. | Three months
  To assess the correlation of EUS-guided portal venous pressure (PVP) and transjugular wedged hepatic venous pressure (WHVP) measurement before treatment start as well as after treatment start with NSBB.
CSPH assessed via EUS-guided pressure measurement. | Three months
  To determine if the current definition of CSPH (i.e. HVPG >/= 10 mmHg) can be adopted for portal tension measurement via EUS-PPG.
Correlation of sequential EUS-PPG and HVPG with non-invasive assessment tools before/after treatment with NSBB. | Three months
  To evaluate the correlation of sequential PPG and HVPG measurements, before and after treatment start with NSBB, with (the evolution of) non-invasive assessment tools. Non-invasive tools evaluated are fibrosis-4 (FIB-4) score, AST to platelet ratio index (APRI), liver stiffness-spleen size-to-platelet ratio-score (LSPS), platelet count to spleen diameter ratio (PSR), liver stiffness measurement (LSM) and spleen stiffness measurement (SSM).
Safety of repeated EUS-PPG | 14 weeks
  To assess the number of participants with any adverse event related to the (repeated) EUS-guided portal pressure gradient measurements. Potential risks associated with the study-specific intervention include fever, (minor) haemorrhage, (minor) infection, inflammation, pain/discomfort, (minor) vessel trauma, vessel occlusion/thrombosis, allergic reaction to medication*, aspiration*, cardiac arrhythmia or arrest*, respiratory depression or arrest*, death*. Adverse events indicated with * are related to the gastrointestinal endoscopic procedure required for the EUS-PPG intervention and are not specific to the device.

CONTACTS AND LOCATIONS:
Overall Officials: Schalk van der Merwe, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospital Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No
Patient confidentiality